CLINICAL TRIAL: NCT01115335
Title: Feasibility, Acceptability, and Safety of Neonatal Male Circumcision at the University Teaching Hospital in Lusaka, Zambia and in the Lusaka District in Zambia Using Gomco; Plastibell; and Mogen Methods
Brief Title: Feasibility, Acceptability, and Safety of Neonatal Male Circumcision in Lusaka, Zambia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University Teaching Hospital, Lusaka, Zambia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PS123541-06
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2010-04

CONDITIONS: Neonatal Male Circumcision
Keywords: neonatal male circumcision; Gomco; Plastibell; Mogen; Safety; Uptake; Acceptability; Feasibility; Zambia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gomco (Active Comparator): NMC performed using a Gomco clamp
  Interventions: Procedure: Neonatal male circumcision
- Mogen clamp (Active Comparator): NMC performed using a Mogen clamp
  Interventions: Procedure: Neonatal male circumcision
- Plastibell (Active Comparator): NMC performed using a Plastibell device
  Interventions: Procedure: Neonatal male circumcision

INTERVENTIONS:
Procedure: Neonatal male circumcision — Circumcision performed on a male infant within the first month of life, using one of 3 devices

SUMMARY:
In this study of neonatal male circumcision (NMC), the investigators will examine acceptability of among parents, feasibility of training providers and implementing services in various clinical settings, and the safety of service provision comparing three different surgical methods: the Gomco; the Plastibell; and the Mogen clamp. This operational study is being conducted to inform the scale up of neonatal male circumcision in Zambia.

DETAILED DESCRIPTION:
As male circumcision becomes one component of Zambia's plan to prevent the spread of HIV, it is important to understand the acceptability, feasibility, and safety of implementing NMC services in various clinical settings.

In this study, we will examine the acceptability of neonatal male circumcision among parents in several ways. First, we will administer a structured questionnaire on NMC to 1000 consenting parents of newborn boys at a tertiary care institution and 1-2 primary care clinics in Lusaka. All parents approached, regardless of whether or not they complete the survey, will also be offered an opportunity to have their sons circumcised. Uptake will be calculated as the percent of parents approached who consent for their sons to be circumcised. Finally, we will assess parental satisfaction with results of the procedure.

To examine the feasibility of training providers and implementing neonatal male circumcision services in various clinical settings, we will train a group of 15-20 health care providers in three different circumcision methods (Gomco clamp, Mogen clamp, and Plastibell) at 2-3 study sites. We will recruit 600 infants to be circumcised during the training. We will use structured questionnaires and skill assessments to evaluate provider competence after completing the training curriculum, provider preferences among the three circumcision methods, and opinion about how NMC should be scaled up within the existing health care system. We will also document logistical difficulties of scaling up NMC services at the study sites.

Finally, we will examine the safety of implementing NMC by collecting and analyzing data on complications resulting from the different circumcision methods.

ELIGIBILITY:
Inclusion Criteria:

* Male infants who are in the first day of life (including infants < 24 hours old) and up to 4 weeks of age will be considered for circumcision
* Gestational age >37 weeks at birth

Exclusion Criteria:

* Any current illness
* Bleeding diathesis or family history of bleeding disorder
* Abnormality of urethra or penile shaft such as hypospadias
* Local infection defined as redness, swelling, or a purulent discharge from the infant penis
* Greater than four weeks of age

Max Age: 28 Days | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 661 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Complication Rate | 0-6 weeks after the circumcision procedure
  Includes intra-operative and post-operative complications such as bleeding, infection, and cosmetic problems

SECONDARY OUTCOMES:
Uptake of NMC | Ongoing, over the course of the study (1.5 years)
  Defined as % of parents of newborn boys approached during recruitment who consent to having their sons cirucumcised
Provider Preferences | Upon completion of training in NMC
  Measure of provider preferences among 3 circumcision devices being compared
Parent Satisfaction | 6 weeks following the circumcision procedure
  Score, between 0 and 100, of each parent's satisfaction with the outcome of the NMC procedure

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Stringer, MD, Principal Investigator — University of Alabama at Birmingham and Centre for Infectious Disease Research of Zambia; Kasonde Bowa, MD, Principal Investigator — University Teaching Hospital, Lusaka, Zambia; John Kachimba, MD, Principal Investigator — University Teaching Hospital, Lusaka, Zambia
Locations (1):
- University Teaching Hospital and Matero Reference Clinic, Lusaka, Zambia

REFERENCES:
- See also: Local NGO in Zambia overseeing study conduct — http://www.cidrz.org/